CLINICAL TRIAL: NCT02890446
Title: A Randomized Control Trial on the Effects of Attentional Focus on Motor Training of the Upper Extremity Using Robotics With Individuals After Chronic Stroke
Brief Title: The Effects of Attentional Focus on Arm Training in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Grace Kim, Assistant Professor, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #1311014488
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
Keywords: attentional focus; upper extremity; hemiparesis; stroke
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Focus (EF) (Experimental): Participants received arm training using the InMotion2 robot under external focus practice conditions and instructions. Participants practiced arm reaching by playing a simple video game.
  EF instructions: "Focus on moving the yellow ball on the screen in a smooth, straight line at a constant speed"; "Move the yellow ball toward the blinking red/orange light"; and "Hit the center of the target and try not to overshoot the target"
  Interventions: Behavioral: upper arm training on the InMotion 2 shoulder robot
- Internal Focus (IF) (Experimental): Participants received arm training using the InMotion2 robot without the video game interface. Participants were instructed to think about how they were moving their arm while completing the arm training tasks.
  IF instructions:
  "think about how you're moving your arm"; "push your arm away from you"; "pull your arm toward you"; "move your arm to the right/left"
  Interventions: Behavioral: upper arm training on the InMotion 2 shoulder robot

INTERVENTIONS:
Behavioral: upper arm training on the InMotion 2 shoulder robot — Both groups practiced shoulder and elbow exercises on a robotic arm device under an external focus or internal focus practice condition.
  Practiced arm reaching in a clock-like design to facilitate horizontal shoulder flexion, extension, abduction, adduction.
  12 sessions--3 times a week for 4 weeks

SUMMARY:
This study compares the effects of an internal versus an external focus of attention on motor training of the affected arm for individuals with stroke. Participants were randomly assigned to either the internal or external focus treatment groups and received 12 sessions of arm training.

DETAILED DESCRIPTION:
Participants were randomized to one of two treatment groups and received upper arm reaching training on the InMotion 2 shoulder robot (12 hourly sessions over four weeks). The external focus group received instructions specifically to pay attention to the task goal--hitting targets on the video game, while the internal focus group was instructed to pay attention to the movement of their arm motions (video game monitor was turned off). Both groups practiced the same arm reaching pattern and were matched for level of arm impairment and training dosage.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke > 6 months
* moderate to severe arm impairment
* intact visual scanning and spatial orientation of the affected arm
* functional cognitive status
* medically stable

Exclusion Criteria:

* concurrent occupational or physical therapy for the arm
* joint contractures at the wrist, forearm, elbow, or shoulder
* moderate to severe spasticity at the elbow or shoulder
* presence of other neurological conditions
* botulinum toxin injection in the affected arm < 3 months prior
* score of 0/5 on manual muscle test at the elbow or shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in coordination at the shoulder and elbow measured by joint independence after arm training assessed start of training, discharge and at follow up. | baseline, 4 weeks, 8 weeks
  kinematic measure of coordination between the shoulder and elbow joint
Change in quality of arm motion measured by smoothness at the start of arm training, at 4week, and 8 weeks. | baseline, 4 weeks, 8 weeks
  kinematic assessment of arm motion measured by average velocity decided by maximum velocity
Change in motor impairment of the arm measured by Fugl-Meyer Assessment (FMA) at the start of training, discharge, and follow up. | baseline, 4 weeks, 8 weeks
  performance based assessment of underlying motor impairment of the affected shoulder, elbow, hand after stroke
Change in motor impairment and functional ability of the arm measured by the Wolf Motor Function Test (WMFT) at start of training, discharge, and follow up. | baseline, 4 weeks, 8 weeks
  performance based assessment of underlying motor impairment and function of the affected arm after stroke

REFERENCES:
- [Background] Kal EC, van der Kamp J, Houdijk H. External attentional focus enhances movement automatization: a comprehensive test of the constrained action hypothesis. Hum Mov Sci. 2013 Aug;32(4):527-39. doi: 10.1016/j.humov.2013.04.001. Epub 2013 Jun 30. PMID 24054892
- [Background] Wulf G, Shea C, Lewthwaite R. Motor skill learning and performance: a review of influential factors. Med Educ. 2010 Jan;44(1):75-84. doi: 10.1111/j.1365-2923.2009.03421.x. PMID 20078758
- [Background] Fasoli SE, Trombly CA, Tickle-Degnen L, Verfaellie MH. Effect of instructions on functional reach in persons with and without cerebrovascular accident. Am J Occup Ther. 2002 Jul-Aug;56(4):380-90. doi: 10.5014/ajot.56.4.380. PMID 12125827
- [Background] Durham KF, Sackley CM, Wright CC, Wing AM, Edwards MG, van Vliet P. Attentional focus of feedback for improving performance of reach-to-grasp after stroke: a randomised crossover study. Physiotherapy. 2014 Jun;100(2):108-15. doi: 10.1016/j.physio.2013.03.004. Epub 2013 Jun 21. PMID 23796803
- [Background] Wulf G, McNevin N, Shea CH. The automaticity of complex motor skill learning as a function of attentional focus. Q J Exp Psychol A. 2001 Nov;54(4):1143-54. doi: 10.1080/713756012. PMID 11765737
- [Derived] Kim GJ, Hinojosa J, Rao AK, Batavia M, O'Dell MW. Randomized Trial on the Effects of Attentional Focus on Motor Training of the Upper Extremity Using Robotics With Individuals After Chronic Stroke. Arch Phys Med Rehabil. 2017 Oct;98(10):1924-1931. doi: 10.1016/j.apmr.2017.06.005. Epub 2017 Jun 24. PMID 28652064